CLINICAL TRIAL: NCT03949842
Title: A Comparison of the Clinical Effectiveness of Inhaled Triple Therapy (Fluticasone Furoate / Umeclidinium Bromide / Vilanterol) in a Single Inhaler (TRELEGY™ ELLIPTA™) With Inhaled Non-ELLIPTA™ Multiple Inhaler Triple Therapies in COPD Patients in the US Within a Usual Care Setting in a Prospective Pre-Post Study
Brief Title: Legend: TRELEGY Real World Chronic Obstructive Pulmonary Disease (COPD) Effectiveness Study
Acronym: LEGEND
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The decision to end the study was based on a change in GSK strategy. No subjects were enrolled into the study.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 206860
Record Dates: First submitted 2019-05-13; First posted 2019-05-14 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Fluticasone furoate; Umeclidinium bromide; Vilanterol; COPD; ELLIPTA; TRELEGY; MITT; SITT
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fluticasone furoate

STUDY DESIGN:
Intervention Model Description: This is a retrospective pre-switch and prospective post-switch study design. Subjects will be on their usual care for the retrospective pre-switch period of the study, then they are enrolled into the study and switched onto Trelegy or FF/UMEC/VI for the prospective period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subjects who inhaled non-ELLIPTA MITT (Experimental): Subjects with moderate or severe exacerbation in the past year and history of use of inhaled non-ELLIPTA MITT of ICS/LABA/LAMA within a routine clinical practice setting in the 52-week retrospective pre-switch period.
  Interventions: Drug: Inhaled corticosteroids/long-acting beta2-adrenergic/long-acting muscarinic receptor antagonists
- Subjects receiving TRELEGY ELLIPTA SITT (Experimental): Subjects will receive FF/UMEC/VI (100 microgram [mcg]/62.5 mcg/25 mcg), inhalation powder, once daily, in a single device (TRELEGY ELLIPTA) in the 52-week prospective post-switch period.
  Interventions: Drug: Fluticasone furoate/umeclidinium/vilanterol

INTERVENTIONS:
Drug: Inhaled corticosteroids/long-acting beta2-adrenergic/long-acting muscarinic receptor antagonists — A fixed dose of combination ICS/LABA plus LAMA once-daily was administered to COPD subjects using two separate non-ELLIPTA devices.
  Arms: Subjects who inhaled non-ELLIPTA MITT
Drug: Fluticasone furoate/umeclidinium/vilanterol — The first strip will contain FF at a dose strength of 100 mcg will be blended with lactose. The second strip will be contain UMEC and VI at a dose strength of 25 mcg and 62.5 mcg blended with lactose and magnesium stearate with respectively.
  Arms: Subjects receiving TRELEGY ELLIPTA SITT

SUMMARY:
The primary purpose of this study is to assess the effectiveness of TRELEGY ELLIPTA single inhaler triple therapy (SITT) (fluticasone furoate/umeclidinium bromide/vilanterol [FF/UMEC/VI]) relative to non-ELLIPTA multiple inhaler triple therapies (MITT) of inhaled corticosteroids/long-acting beta2-adrenergic receptor agonists/muscarinic receptor antagonists (ICS/LABA/LAMA) within a routine clinical practice setting. This is a non-randomized, interventional and self-controlled cohort study conducted to collect data in routine practice. This study will have two periods where in retrospective data will be collected in pre-switch period and prospective data will be collected in post-switch periods. Subjects will be switched from non-ELLIPTA MITT to TRELEGY ELLIPTA. The pre-switch period is of 52 weeks and post-switch period will be of 52 weeks. Additionally subjects will receive safety follow-up call at 26 weeks and 52 weeks for safety monitoring. Approximately 1300 subjects will be enrolled for this study. TRELEGY ELLIPTA is a registered trademark of the GlaxoSmithKline (GSK) group of companies.

ELIGIBILITY:
Inclusion Criteria

* Subject must be at least 40 years of age at the time of signing the informed consent.
* Subjects with a documented physician diagnosis of COPD.
* Subjects who have been prescribed non-ELLIPTA MITT for daily use for at least 52 weeks prior to Visit 1.
* Male and/or female. Female subjects: A female subject is eligible to participate if she is not pregnant, not breastfeeding, and not a woman of childbearing potential.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).

Exclusion Criteria

* Women who are: Pregnant or lactating or are planning on becoming pregnant during the study and of child bearing potential.
* Subjects with an exacerbation with an onset within 4 weeks before Visit 1 must not be enrolled. Enrollment should be delayed until at least 4 weeks after the onset of an exacerbation or until the exacerbation has resolved, whichever is the longer.
* Subjects with any life threatening condition (low probability in the opinion of the Investigator of 52 weeks survival due to severity of COPD or co-morbid condition at Visit 1.
* Subjects with historical or current evidence of uncontrolled or clinically significant disease. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the subject at risk through participation, or which would affect the effectiveness or safety analysis if the disease/condition exacerbated during the study.
* Subjects with severe milk-protein allergy or who have demonstrated hypersensitivity to FF/UMEC/VI or any of the excipients in TRELEGY ELLIPTA.
* Subjects currently participating in any other study.
* Subjects taking any investigational drug treatment within 30 days prior to Visit 1 or within five half-lives (t1/2) of completion of the prior investigational study (whichever is the longer of the two).
* Subjects who are planning or may plan to change health plan or physician/investigator during the 52-week study.
* Subjects who, in the opinion of the treating physician, are considered to be a chronic user of oral corticosteroids (including oral and injectable) for respiratory or other indication in the past 52 weeks (if unsure discuss with the medical monitor prior to screening).
* Subjects who have received a course of systemic corticosteroids for reasons other than COPD exacerbations within the 4 weeks prior to Visit 1.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of moderate, severe COPD exacerbations | 104 weeks
  Moderate and severe COPD exacerbations will be defined using an algorithm agreed upon by GlaxoSmithKline and the health plans that identifies these events from health plan medical claims data. Moderate exacerbation is any physician office visit, urgent care visit or emergency room visit for COPD where any oral corticosteroids or antibiotics are prescribed during visit. Severe exacerbations are any COPD related inpatient visit. Exacerbations will be determined in the same fashion in the retrospective pre-switch period and the prospective post switch period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Waterbury, Connecticut
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Layton, Utah

IPD SHARING:
Plan to Share IPD: No